CLINICAL TRIAL: NCT03442881
Title: The Use of International Ovarian Tumor Analysis and Assessment of Different Neoplasia in the Adnexa Model in Differentiating Malignant and Benign Adnexal Masses
Brief Title: The Use of International Ovarian Tumor Analysis and Assessment of Adnexal Neoplasia in Differentiating Malignant and Benign Adnexal Masses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Other Study IDs: 28
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Adnexal Mass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- benign adnexal mass: pathological examination of the specimen after excision reveals benign criteria
  Interventions: Procedure: Excision of adnexal mass through laprotomy
- Malignant adnexal mass: pathological examination of the specimen after excision reveals malignant criteria
  Interventions: Procedure: Excision of adnexal mass through laprotomy

INTERVENTIONS:
Procedure: Excision of adnexal mass through laprotomy — Through laparotomy incision, the adnexal mass will be excised

SUMMARY:
All participants will be subjected to Serum measurements of CA-125 by the immunoradiometric assay, Ultrasound evaluation of the Adnexal masses which is described according to origin (ovarian/extraovarian); position (right/left/bilateral); number of lesions; type of lesions (unilocular/multilocular); size in three dimensions (longitudinal, anteroposterior and transverse diameters); intracystic fluid echogenicity; number of loculations; presence and size of septations (only thickest one of septations is considered); presence, number and size of solid papillary projections (largest thickness is considered); presence and size of the largest solid component (three diameters); presence and measurement of fluid volume in the posterior cul-de-sac and presence and location of lesions suggestive of metastases. Then surgical intervention will be done with pathological examination of the specimen

DETAILED DESCRIPTION:
All participants will be subjected to Serum measurements of CA-125 by the immunoradiometric assay, Ultrasound evaluation of the Adnexal masses which is described according to origin (ovarian/extraovarian); position (right/left/bilateral); number of lesions; type of lesions (unilocular/multilocular); size in three dimensions (longitudinal, anteroposterior and transverse diameters); intracystic fluid echogenicity; number of loculations; presence and size of septations (only thickest one of septations is considered); presence, number and size of solid papillary projections (largest thickness is considered); presence and size of the largest solid component (three diameters); presence and measurement of fluid volume in the posterior cul-de-sac and presence and location of lesions suggestive of metastases. Then surgical intervention will be done with pathological examination of the specimen

ELIGIBILITY:
Inclusion Criteria:

* Women with clinically and sonographically diagnosed adenxal mass more than 5 cm in diameter. 2. Patients who will undergo surgical intervention . 3. Patients are recruited regardless of age, parity and complaint

Exclusion Criteria:

* Patients treated with conservative management. 2. Patients known to be pregnant.

Ages: 15 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study included 80 patients who had a preliminary diagnosis of adnexal mass clinically and/or sonographically
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Nature of the mass | At time of surgery
  Benign or malignant criteria of the excised adnexal mass

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt